CLINICAL TRIAL: NCT00095069
Title: A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel-Groups Efficacy and Safety Extension Study of MK0928 in the Treatment of Adult Outpatients With Primary Insomnia
Brief Title: Efficacy and Safety of MK0928 for Insomnia in Adults (0928-003)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-003; MK0928-003; 2004_086
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0928, gaboxadol / Duration of Treatment - 1 year
Drug: Comparator: placebo / Duration of Treatment -1 year

SUMMARY:
The purpose of this trial is to study the safety and effectiveness of MK0928 for adults with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600
Dates: Start 2004-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Patient-reported amount of sleep and time to fall sleep at night after three months

SECONDARY OUTCOMES:
Patient-reported awakenings at night
Sleep quality
Functioning after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Roth T, Lines C, Vandormael K, Ceesay P, Anderson D, Snavely D. Effect of gaboxadol on patient-reported measures of sleep and waking function in patients with Primary Insomnia: results from two randomized, controlled, 3-month studies. J Clin Sleep Med. 2010 Feb 15;6(1):30-9. PMID 20191935